CLINICAL TRIAL: NCT02146235
Title: The Effects of Music Therapy in the Treatment of Chronic Obstructive Pulmonary Disease
Brief Title: Music Therapy in the Treatment of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 081-08
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Diseases
Keywords: Music Therapy; Pulmonary Disease; COPD; Music Visualization; Therapeutic Singing; Wind-playing; Lung Condition
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group - Music Therapy (Experimental): The experimental group participates in once weekly group music therapy session for 6 weeks using playing of simple wind instruments, singing, and music visualization. The Music therapy session lasts 45 min. and encourages patients to use breathing techniques to achieve a relaxation response. Extructured techniques involving singing, music improvisation supports breath pattens and provides supporting coping styles. The use of wind instruments involves a focus of breathing efficiently and elongating the exhalation to prolong musical tones and transferring breath control. Music Visualization involving deep breathing techniques provides optimal mind-body connection, influences breathing rhythms through more indirect means while reducing stress, accessing altered states and encourages healing imagery.
  Interventions: Behavioral: Psycho-Music Therapy
- Standard Pulmonary Rehabilitation (No Intervention): Pulmonary rehabilitation is a program to people with chronic lung diseases like COPD, emphysema, and chronic bronchitis lead full, satisfying lives and restore them to their highest functional capacity. Pulmonary rehab is aimed to improve quality of life by:
  Decreasing respiratory symptoms and complications Encouraging self-management and control over daily functioning Improving physical conditioning and exercise performance Improving emotional well-being Reducing hospitalizations
  Pulmonary rehab programs include:
  Medical management Exercise Breathing retraining Education Emotional support Nutrition counseling

INTERVENTIONS:
Behavioral: Psycho-Music Therapy
  Arms: Treatment Group - Music Therapy

SUMMARY:
The investigators combine traditional medical care with an integrative modality - Music Therapy specifically including wind playing, singing, and music visualizations- to study the effects on physical function and quality of life for adults with COPD. The primary goals are to increase respiratory function and reduce respiratory symptoms and hospitalizations in order to improve breathing, functional capacity for activities of daily living, psychological well-being and quality of life in adult age 45 and above who are diagnosed with COPD

DETAILED DESCRIPTION:
This study examines the effect of a multimodal psycho-music therapy intervention on respiratory symptoms (dyspnea), depression, and quality of life of patients with pulmonary disease during Pumonary Rehabilitation, in the combined effort of two departments of Mount Sinai Beth Israel: The Alice Lawrence Center for Health and Rehabilitation and The Louis Armstrong Center for Music and Medicine

1. Desing The study cohort included patient with at least moderate COPD according to the GOLD classification as well as other chronic disabling respiratory diseases. Inclusion criteria were defined as being enrolled in a Pulmonary Rehabilitation (PR) program as well as the ability to attend music therapy sessions at least once a week for 5 of 6 weekly sessions. The patients were required to be medically stable simultaneously allowing them to participate in the pulmonary rehabilitation program. Standard, routine pulmonary rehabilitative medical care was used as the control to music therapy plus PR and patient selection was provided by a computer generated randomization protocol. The intervention included live music listening with visualization, wind playing and singing undertaken to study their effects on perceived dyspnea, depression and quality of life. Patients were allowed to choose between easy to play wind instruments i.e recorder, slide whistle, harmonica, etc. and instructed on their use. Ninety- eight subjects were evaluated as potential candidates for the study. Thirty of them were excluded because they would not commit to participate in the required number of music therapy sessions either due to the anticipated time commitment or personal/medical concerns. The 68 patients who agreed to participate in the investigation (Age Mean: 70.1), were randomize and 38 were allocated to the treatment group and 30 to the control group. These 68 patients who were newly enrolled in the Alice Lawrence Center had voluntarily sought to participate active PR through advertising and flyers posted in the community and throughout the hospital and affiliated office practices. The weekly music therapy sessions lasted 45 min, for a period of 6 weeks, in groups of 6 participants or less.

2- Method At the beginning and end of each session the patients were asked to score the intensity of current breathlessness by drawing a circle on different pictures of lungs that represented extent of dyspnea (VAS) These recorded measures would be collected at the end of each session, in order to evaluate the subjective effect of the treatment on the patients perception of dyspnea. CRQ and BDI were also administered at the beginning of the PR program and subsequently at 6 weeks, the end of the PR program. In the music therapy group, every session included music visualizations, wind instrument playing, and singing, providing direct methods of working with the breath control and offering active music-making experiences to support optimal breathing, foster self-expression, and increase opportunities for coping with the challenges of chronic respiratory disease.

3-Outcome measures

Primary outcomes were depressive symptoms, disease-specific quality of life factors, and patients' perceived dyspnea:

* Depressive symptoms were evaluated using the Beck Depression Inventory 2nd edition-Fast Screen (BDI-FS), a 7-item subscale of the BDI-II. The BDI-FS measures signs and symptoms such as sadness, pessimism, past failure, anhedonia, self-dislike, self-criticalness, and suicidal thoughts or ideation.
* Disease-specific quality of life as measured by the Chronic Respiratory Questionnaire Self-Reported (CRQ-SR) is divided into four dimensions of dyspnea, fatigue, emotional function and mastery, with a 7-point Likert scale response for each question. Dyspnea relates to a patient's symptoms of shortness of breath and difficulty breathing. Mastery relates to a patient's sense of having control over his or her disease and symptoms. Emotion relates to a patient's general mood. Fatigue relates to a patient's energy level. We measured CRQ-SR domain scores at the time of enrolment in the study and again at completion, immediately following the final session after six weeks).
* Visual Analogue Scale (VAS) scale. This measures perceived dyspnea or breathlessness in participants during the music therapy sessions. The VAS is widely used in the measurement of breathlessness as well as other symptoms, e.g. pain, anxiety (annotate to appendix)

  4-Statistical analysis Each of the dependent measures of primary outcomes (Depression, Dyspnea, and Health-Related Quality of Life) was analyzed using a generalized linear mixed model (SAS Proc GLIMMIX, SAS 9.3) involving a single between subjects factor (Treatment vs. Control) and a single within subjects factor (Period - enrollment vs. follow up 6 weeks later) Test of Treatment Group differences at Enrollment and at 6 weeks were made using planned contrast on the Least-Square means.

ELIGIBILITY:
Inclusion Criteria:

* Patient with at least moderate COPD according to the GOLD classification as well as other chronic disabling respiratory diseases. Inclusion criteria were defined as being enrolled in a Pulmonary Rehabilitation (PR) program as well as the ability to attend music therapy sessions at least once a week for 5 of 6 weekly sessions.
* The patients were required to be medically stable simultaneously allowing them to participate in the pulmonary rehabilitation program

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Chronic Respiratory Questionnaire Self-Reported (CRQ-SR) | up to six weeks
  CRQ-SR is divided into four dimensions of dyspnea, fatigue, emotional function and mastery, with a 7-point Likert scale response for each question. Dyspnea relates to a patient's symptoms of shortness of breath and difficulty breathing. Mastery relates to a patient's sense of having control over his or her disease and symptoms. Emotion relates to a patient's general mood. Fatigue relates to a patient's energy level. Patients generally report that they feel better with an average improvement of 0.5 per dimension. Changes between 0.75 and 1.25 represent important changes of moderate magnitude, and changes greater than 1.5 represent important changes of large magnitude.
Beck Depression Inventory 2nd edition-Fast Screen (BDI-FS) | up to six weeks
  BDI-FS), a 7-item subscale of the BDI-II. The BDI-FS measures signs and symptoms such as sadness, pessimism, past failure, anhedonia, self-dislike, self-criticalness, and suicidal thoughts or ideation. (P5:22). Each question on the BDI is answered on a scale of 0-3 (zero being little or none, and 3 representing a high level of the characteristic in question). Therefore the scale for the sum of the 7 questions goes from 0-21. The suggested scoring is 0-3 = minimal symptoms of depression, 4-6 = mild symptoms of depression, 7-9 = moderate symptoms of depression, and 10-21 = severe symptoms of depression.
Perceived dyspnea Visual Analogue Scale (VAS) | Treatment group only. It is administrated prior and post every music therapy session. (6 weeks)
  A visual analogue scale, consisted in a succession of lung draws representing the breathlessness process with a numerical rating scale. This unidimensional instrument is commonly used in the measurement of dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States

REFERENCES:
- [Background] Bauldoff GS, Rittinger M, Nelson T, Doehrel J, Diaz PT. Feasibility of distractive auditory stimuli on upper extremity training in persons with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2005 Jan-Feb;25(1):50-5. doi: 10.1097/00008483-200501000-00011. PMID 15714113
- [Background] Panigrahi A, Sohani S, Amadi C, Joshi A. Role of music in the management of chronic obstructive pulmonary disease (COPD): a literature review. Technol Health Care. 2014;22(1):53-61. doi: 10.3233/THC-130773. PMID 24398814
- [Background] Bauldoff GS, Hoffman LA, Zullo TG, Sciurba FC. Exercise maintenance following pulmonary rehabilitation: effect of distractive stimuli. Chest. 2002 Sep;122(3):948-54. doi: 10.1378/chest.122.3.948. PMID 12226037
- [Background] von Leupoldt A, Taube K, Schubert-Heukeshoven S, Magnussen H, Dahme B. Distractive auditory stimuli reduce the unpleasantness of dyspnea during exercise in patients with COPD. Chest. 2007 Nov;132(5):1506-12. doi: 10.1378/chest.07-1245. Epub 2007 Sep 21. PMID 17890458
- [Background] Pfister T, Berrol C, Caplan C. Effects of music on exercise and perceived symptoms in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 1998 May-Jun;18(3):228-32. doi: 10.1097/00008483-199805000-00007. PMID 9632325
- [Background] Thornby MA, Haas F, Axen K. Effect of distractive auditory stimuli on exercise tolerance in patients with COPD. Chest. 1995 May;107(5):1213-7. doi: 10.1378/chest.107.5.1213. PMID 7750308
- [Background] Ho CF, Maa SH, Shyu YI, Lai YT, Hung TC, Chen HC. Effectiveness of paced walking to music at home for patients with COPD. COPD. 2012 Aug;9(5):447-57. doi: 10.3109/15412555.2012.685664. Epub 2012 May 29. PMID 22643033
- [Background] Louie SW. The effects of guided imagery relaxation in people with COPD. Occup Ther Int. 2004;11(3):145-59. doi: 10.1002/oti.203. PMID 15297895
- [Background] Singh VP, Rao V, V P, R C S, K KP. Comparison of the effectiveness of music and progressive muscle relaxation for anxiety in COPD--A randomized controlled pilot study. Chron Respir Dis. 2009;6(4):209-16. doi: 10.1177/1479972309346754. PMID 19858350
- [Background] le Roux FH, Bouic PJ, Bester MM. The effect of Bach's magnificat on emotions, immune, and endocrine parameters during physiotherapy treatment of patients with infectious lung conditions. J Music Ther. 2007 Summer;44(2):156-68. doi: 10.1093/jmt/44.2.156. PMID 17484523
- [Background] Sliwka A, Nowobilski R, Polczyk R, Nizankowska-Mogilnicka E, Szczeklik A. Mild asthmatics benefit from music therapy. J Asthma. 2012 May;49(4):401-8. doi: 10.3109/02770903.2012.663031. Epub 2012 Mar 7. PMID 22397390
- [Background] Muller V, Lindenberger U. Cardiac and respiratory patterns synchronize between persons during choir singing. PLoS One. 2011;6(9):e24893. doi: 10.1371/journal.pone.0024893. Epub 2011 Sep 21. PMID 21957466
- [Background] Irons JY, Kenny DT, Chang AB. Singing for children and adults with bronchiectasis. Cochrane Database Syst Rev. 2010 Feb 17;2010(2):CD007729. doi: 10.1002/14651858.CD007729.pub2. PMID 20166097
- [Background] Herer B. [Outcomes of a pulmonary rehabilitation program including singing training]. Rev Mal Respir. 2013 Mar;30(3):194-202. doi: 10.1016/j.rmr.2012.10.602. Epub 2012 Dec 13. French. PMID 23497929
- [Background] Lord VM, Hume VJ, Kelly JL, Cave P, Silver J, Waldman M, White C, Smith C, Tanner R, Sanchez M, Man WD, Polkey MI, Hopkinson NS. Singing classes for chronic obstructive pulmonary disease: a randomized controlled trial. BMC Pulm Med. 2012 Nov 13;12:69. doi: 10.1186/1471-2466-12-69. PMID 23145504
- [Background] Bonilha AG, Onofre F, Vieira ML, Prado MY, Martinez JA. Effects of singing classes on pulmonary function and quality of life of COPD patients. Int J Chron Obstruct Pulmon Dis. 2009;4:1-8. Epub 2009 Apr 15. PMID 19436683
- [Background] Goodridge D, Nicol JJ, Horvey KJ, Butcher S. Therapeutic Singing as an Adjunct for Pulmonary Rehabilitation Participants With COPD Outcomes of a Feasibility Study. Music and Medicine 2013; 5(3): 169-176.
- [Background] BOUHUYS A. LUNG VOLUMES AND BREATHING PATTERNS IN WIND-INSTRUMENT PLAYERS. J Appl Physiol. 1964 Sep;19:967-75. doi: 10.1152/jappl.1964.19.5.967. No abstract available. PMID 14207753
- [Background] Bouhuys A (1968) Pressure-flow events during wind instrument playing. Ann New York Acad Sci 155(1):264-275
- [Background] Zuskin E, Mustajbegovic J, Schachter EN, Kern J, Vitale K, Pucarin-Cvetkovic J, Chiarelli A, Milosevic M, Jelinic JD. Respiratory function in wind instrument players. Med Lav. 2009 Mar-Apr;100(2):133-41. PMID 19382523
- [Background] Alexander JL, Wagner CL. Is harmonica playing an effective adjunct therapy to pulmonary rehabilitation? Rehabil Nurs. 2012 Jul-Aug;37(4):207-12. doi: 10.1002/rnj.33. Epub 2012 Jun 18. PMID 22744994
- [Background] Bausewein C, Booth S, Gysels M, Higginson IJ. WITHDRAWN: Non-pharmacological interventions for breathlessness in advanced stages of malignant and non-malignant diseases. Cochrane Database Syst Rev. 2013 Nov 22;2013(11):CD005623. doi: 10.1002/14651858.CD005623.pub3. PMID 24272974